CLINICAL TRIAL: NCT04486339
Title: Pulmonary Vein Isolation Using Stereotactic Radiotherapy System for the Treatment of Refractory Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2019-047-4
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stereotactic body radiotherapy (SBRT) (Experimental): Noninvasive SBRT will be delivered in a single fraction to electrical isolate the pulmonary veins under CT-guidance.
  Interventions: Radiation: Stereotactic Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Radiotherapy — Stereotactic radiotherapy targets on the pulmonary vein ostium aiming to achieve pulmonary vein electrial isolation

SUMMARY:
The study aims to investigate the short-term (3 months) and intermediate-term (12 months) safety and preliminary efficacy of stereotactic radiotherapy for pulmonary vein isolation to treat refractory atrial fibrillation.

DETAILED DESCRIPTION:
This is a single center, single arm, prospective and phase 1 clinical trial. Patients with refractory atrial fibrillation (AF) will receive single fraction stereotactic radiotherapy for pulmonary vein isolation. To minimize the potential risks associated with this innovative technique, the study has been designed in a stepwise dose escalation fashion under carefully observation by the investigators. The dose escalation is guided by 3+3 algorithm to ensure more patients will be spared dose limiting toxicities and more patients will be entered on the dose level than will be chosen as optimal dose of maximal effects. Low dosing levels with established safety profile will first be applied before administering higher dosing levels based on preclinical studies.

Safety is the primary endpoint of the study. Safety will be assessed by incidence and evaluation of any serious adverse evens using CTCAE V5.0 criteria associated with the procedure through 90 days (short-term) and 12 months (intermediate term). Efficacy will be evaluated by assessing atrial fibrillation recurrence (for paroxysmal AF) or AF burden (for persistent AF) after 90 days of blank period until 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

Paroxysmal or persistent atrial fibrillation. Age 55-89 Symptomatic, refractory to at least 3 antiarrhythmic drugs Failure from the previous catheter ablation of atrial fibrillation, or contraindicate /unwilling to undergo catheter ablation.

Anticoagulation for at least 3 months if CHA2DS2-VASc 2 or more.

Exclusion Criteria:

With concomitant atrial flutter, WPW syndrome or supraventricular tachycardia. With sustained ventricular tachycardia. With sick sinus syndrome or atrioventricular block fulfilling the indication of permanent pacemaker implantation.

Stroke or myocardial infarction within 8 weeks. Uncontrolled heart failure or unstable angina pectoris. Severe structral heart diseases. Severe pulmonary hypertension. Uncontrolled hypertension. Severe respiratory disease. Esophageal ulcer. Intracardiac thrombus by TEE. Pregnancy or have a preganancy plan. Others.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
90 days adverse events by CTCA5 | 90 days
  Safety will be assessed by incidence and evaluation of any adverse events using CTCA5 V5.0 criteria that are related to the procedure

SECONDARY OUTCOMES:
12 months adverse events by CTCA5 | 12 months
  Safety will be assessed by incidence and evaluation of any adverse events using CTCA5 V5.0 criteria that are related to the procedure
Recurrence of atrial fibrillation (for paroxysmal atrial fibrillation) | 90 days to 12 months
  Recurrence of atrial fibrillation after 90 days blanking period post-treatment
Atrial fibrillation burden reduction (for persistent atrial fibrillation) | 90 days to 12 months
  Atrial fibriilation burden reduction after 90 days blanking period post-treatment
All-cause motality | 12 months
  Motality due to any reason
Quality of life improvement | 3 month, 6 month and 12 month
  Quality of life after the procedure evaluated by the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Gang Li, Principal Investigator — Xinhua Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Xinhua Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China